CLINICAL TRIAL: NCT04777825
Title: Evaluation of the Effectiveness of a Heart Rate Variability Biofeedback Training in the Management of Dysfunctional (Somatoform) Disorders
Brief Title: Heart Rate Variability Biofeedback Training in Psychogenic Disorders
Acronym: ECoDys
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL19_0346
Record Dates: First submitted 2020-09-08; First posted 2021-03-02 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Psychogenic Dystonia
Keywords: Cervical dystonia; Psychogenic disorder; Heart Rate Variability; Functional neurosurgery
MeSH Terms: conditions — Dystonic Disorders; Torticollis; Somatoform Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HRV biofeedback training (Experimental): During the inclusion visit, all patients will benefit from a psychoeducation session supervised by the psychologist. This group of patients will also benefit from the HRV biofeedback training.
  Interventions: Other: Heart rate variability biofeedback training (Symbiocenter); Other: psychoeducation session
- control (Other): During the inclusion visit, all patients will benefit from a psychoeducation session supervised by the psychologist.
  Interventions: Other: psychoeducation session

INTERVENTIONS:
Other: Heart rate variability biofeedback training (Symbiocenter) — 12 sessions of thirty minutes. Patients will participate through several serious game associated with HRV biofeedback training
  Arms: HRV biofeedback training
Other: psychoeducation session — Each patient will therefore be presented individually with a Powerpoint consisting of 35 slides divided into 4 sub-sections explaining in a fun and educational format the physiological model of stress, the respiratory function and its benefits, presentation of various relaxation techniques and recommendations for reading (stress management, letting go, mindfulness meditation) and other tools to help relaxation (smartphone applications).

SUMMARY:
To study whether Heart Rate Variability (HRV) biofeedback training can improve abnormal head posture and painful symptomatology in patients with "cervical dystonia" not selected for DBS after extensive screening in a specialized unit but diagnosed " dysfunctional ".

Patients of the respiratory coherence group will receive HRV biofeedback training for 12 sessions during a 6 months-period. The hypothesis is that this kind of physiological noninvasive therapy increasing coherence respiratory, will reduce pain and patient's complain about their psychogenic abnormal head posture. Improvement of anxiety, depression and quality of life are expected.

DETAILED DESCRIPTION:
Patients presenting with an isolated abnormal head posture, first diagnosed as cervical dystonia, demonstrated in fact, after neurological screening, to be of psychogenic origine. These patients are not candidate for functional surgery and, furthermore, usually refuse psychotherapy leading them to medical nomadism. This study proposes to evaluate the efficacy of an innovative intervention program based on Heart Rate Variability (HRV) biofeedback that promotes self-regulatory skills in dysfunctional movement disorders (DMD) patients in order to improve their condition and symptomatology.

Heart rate is under the control of efferent sympathetic and vagal activities directed to the sinus node, which are modulated by central brain stem (vasomotor and respiratory centers) and peripheral oscillators (oscillation in arterial pressure and respiratory movements). Spectral analysis of HRV is a reliable quantitative method for analyzing the modulatory effects of neural mechanisms on the sinus node. Several biofeedback protocols and assistive electronic technologies, such as proposed by SymbioCenter©, exist to enhance increase HRV and synchronize respiration with the heart rhythm. HRV biofeedback training appears to be an opportunity in the patient's management in order of preventing medical overconsuming. It is offering a safe and non-pharmacological alternative approach managed by a multidisciplinary team in a functional neurosurgery unit. It is expected that developing respiratory coherence in these patients will improve their painful symptomatology.

ELIGIBILITY:
Inclusion criteria:

* Age 18 to 75
* Responding to somatoform disorder characteristics as described in ICD-10 (F45: "The onset of physical symptoms associated with an insistent medical quest, persisting despite repeated negative assessments and statements by physicians that the symptoms have no organic basis. If there is a genuine physical disorder, it does not account for the nature or severity of the symptoms, or the distress or concerns of the subject. The multidisciplinary team will determine whether or not the diagnosis of conversion disorder (disorder with functional neurological symptoms) of the DSMV (300.11) [ICD-10 equivalent: F44.4 "dissociative disorder with abnormal movements"] is associated with the diagnosis of conversion disorder (disorder with functional neurological symptoms) of the DSMV (300.11) [ICD-10 equivalent: F44.4 "dissociative disorder with abnormal movements"], selected by the multidisciplinary team after a phase 1 assessment.
* Patient benefiting from a social security scheme

Exclusion criteria:

* Simulation identified with obvious search for secondary benefit according to the ICD-10 classification ( Z76.5 Simulator: Person pretending to be ill (with obvious motivation"), or DSM-V(V65.2)
* Any other specific PAT-specific CEP (botulinum toxin, psychotherapy and/or relaxation provided by a professional (CBT, ACT, Mindfulness, etc.)) scheduled within 6 months, with the exception of the usual analgesics (Tier I or II)Presenting significant cognitive impairment (MoCa test ≤ 24/30),
* Absence foreseeable at least 30% of the sessions,
* Lack of informed consent.
* Pregnancy or planned pregnancy during the study period, Pregnant or breastfeeding women
* Major protected by law or patient under guardianship or curatorship
* Participation in other ongoing research

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Variability of the cervical dystonia at 6 months | 6 months
  Measured by the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) scale. The total score is 0 (better outcome) to 85 (worse outcome)

SECONDARY OUTCOMES:
Variability of the cervical dystonia at 3 months | 3 months
  Measured by the Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) scale. The total score is 0 (better outcome) to 85 (worse outcome)
Quality of life assessment in cervical dystonia at 3 months | 3 months
  Measured by the Craniocervical Dystonia Questionnaire (CDQ24) scale
Quality of life assessment in cervical dystonia at 6 months | 6 months
  Measured by the Craniocervical Dystonia Questionnaire (CDQ24) scale
Quality of life assessment at 3 months | 3 months
  Measured by SF-36 scale
Quality of life assessment at 6 months | 6 months
  Measured by SF-36 scale
Assessment of the severity of depression at 3 month | 3 months
  Measured by Beck Depression Inventory (BDI-II) scale
Assessment of the severity of depression at 6 month | 6 months
  Measured by the Beck Depression Inventory (BDI-II) scale
Assessment of the anxiety at 3 month | 3 months
  Measured by the State-Trait Anxiety Inventory (STAI A & B) scale
Assessment of the anxiety at 6 month | 6 months
  Measured by the State-Trait Anxiety Inventory (STAI A & B) scale
satisfaction with the care | 6 months
  satisfaction's VAS
medical nomadism index | 6 months
  The index of "presumed nomadism" is the difference between the number of different doctors consulted and the number of different specialties of these same doctors. Any patient whose index is ≥ 3 over a period of 6 months is presumed nomadic.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe COUBES, MD, PhD, Principal Investigator — Montpellier University Hospital
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No